CLINICAL TRIAL: NCT07222228
Title: A Phase 2b Study to Evaluate the Efficacy and Safety of Subcutaneous Levonorgestrel Butanoate for Female Contraception
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous Levonorgestrel Butanoate for Female Contraception
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Clint Dart, Senior Program Director, NICHD, Premier Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCN021B
Record Dates: First submitted 2025-10-22; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Healthy Women; Female Contraception
Keywords: Female contraception
MeSH Terms: interventions — levonorgestrel butanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LB 60 mg SQ (70 mg/mL) (Experimental): The participants will receive 2 injections of LB 60 mg SQ (70 mg/mL); 1 at Visit 2 (Day 1) and 1 at Visit 7 (Day 120).
  Interventions: Drug: Levonorgestrel butanoate

INTERVENTIONS:
Drug: Levonorgestrel butanoate — 60 mg SQ (70 mg/mL)
  Other Names: Chemical, Generic: 13β-ethyl-17α-ethynylgon-4-en-3-one- 17β-n-butyrate; Trade Names: CDB-1830 and HRP002

SUMMARY:
This is a multicenter, open-label, Phase 2b study to evaluate the efficacy and safety of 2 LB SQ injections administered at a 4-month (approximately 17 weeks) interval for female contraception.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 2b study to evaluate the efficacy and safety of 2 LB SQ injections administered at a 4-month (approximately 17 weeks) interval for female contraception. The study plans to enroll approximately 165 female participants, 18 to 35 years of age, inclusive, at enrollment (Visit 2, Day 1), who have good general overall health. They also must have menstrual cycles of 21 to 35 days when not using hormonal contraception with typical variation in cycle length of 5 days or less, have an intact uterus and at least 1 ovary, expect to have heterosexual intercourse at least once per month during the study, and agree to use no additional methods of contraception during the study. Participants will be excluded if they are planning pregnancy during study participation through the End-of-Treatment Visit (Visit 11, Day 240). In addition, participants must have had 2 spontaneous menses (1 cycle) since delivery, 1 menses following first or second trimester abortion or miscarriage, must not be breastfeeding, or be within 30 days of discontinuing breastfeeding unless the participant has already had 1 cycle (2 menses) following discontinuation of breastfeeding.

The primary aim of the study is to evaluate the contraceptive efficacy of LB SQ injections over 8 cycles. Additionally, LB safety will be assessed based on the incidence of AEs (including weight increase) and injection site reactions and changes from baseline laboratory parameters. The number of bleeding and spotting days per 30-, 90-, and 120-day intervals, as well as responses from the acceptability and satisfaction questionnaire at Day 240 (Month 8), are also secondary endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant understands and signs an ICF approved by the institutional review board prior to any screening activities.
2. Female and 18 to 35 years of age, inclusive, at enrollment (Visit 2, Day 1).
3. Good general overall health with no chronic medical conditions that result in periodic exacerbations requiring significant medical care.
4. Menstrual cycles of 21 to 35 days in length with typical variation in cycle length of 5 days or less when not using hormonal contraception.
5. Intact uterus and at least 1 ovary.
6. If used a hormonal contraceptive or intra-uterine device (IUD) prior to enrollment, the participant meets the appropriate criteria for time since last use:

   1. Oral, transdermal, vaginal, copper or LNG IUD or implantable hormonal contraceptives: participants must have discontinued hormone use ≥4 days prior to start of study treatment, experienced bleeding that is consistent with menses in the opinion of the investigator and not have had unprotected intercourse since discontinuing the method.
   2. Injectable contraception (e.g., DMPA): No injection during the 10 months prior to the Screening Visit, unless the participant has returned to normal menses (i.e., 2 consecutive menses) since last injection.
7. Negative urine pregnancy test at enrollment (Visit 2, Day 1).
8. Body mass index <40 kg/m2.
9. Willing to use the study method as the primary method of contraception until the end of the Treatment Period.
10. At risk for pregnancy defined as:

    1. Expecting to have ≥1 act of heterosexual intercourse each month during study participation until the end of the Treatment Period.
    2. No medical history suggesting possible infertility or hypofertility, including but not limited to, ectopic pregnancy or pelvic infection (unless has had a subsequent intra-uterine pregnancy).
    3. Has a sexual partner with no known problems with infertility orhypofertility.

Exclusion Criteria:

1. Planning pregnancy during study participation through the End -of -Treatment Visit (Visit 11, Day 240).
2. Is post-partum and has not had 2 spontaneous menses (1 cycle) since delivery or 1 menses since first or second trimester abortion or miscarriage.
3. Breastfeeding or within 30 days of discontinuing breastfeeding unless the participant has already had 2 menses (1 cycle) following discontinuation of breastfeeding.
4. Undiagnosed abnormal genital bleeding.
5. Undiagnosed vaginal discharge, lesions, or abnormalities.
6. Participating in another clinical study involving an IP or device within 30 days prior to the Screening Visit or planning to participate in another clinical study during this study.
7. Not living in the catchment area of the study site.
8. Known hypersensitivity or contraindication to progestins, including the active substance LB or any excipients of the study treatment.
9. Current need for therapeutic anticoagulation or known history of thrombophilia.
10. Use or planned use of exogenous reproductive hormones during study participation.
11. Body weight change exceeding 10% over the previous year or planned significant weight loss during the study related to bariatric surgery, dieting, or planned treatment.
12. Uncontrolled hypertension, in which diastolic blood pressure remains ≥95 mmHg or systolic blood pressure remains ≥145 mmHg.
13. Smoking nicotine (e.g., cigarettes or electronic cigarettes) AND has at least 1 of the following comorbidities or conditions (at the discretion of the investigator):

    * Current or history of venous thrombophlebitis or thromboembolic disorders (including deep vein thrombosis and pulmonary embolism).
    * Current or history of cerebrovascular or coronary-artery disease.
    * Valvular heart disease with thrombogenic complications.
    * Diabetes with vascular involvement.
    * Known inherited or acquired predisposition to venous thromboembolism or arterial thromboembolism (e.g., factor VLeiden, prothrombin mutation, antiphospholipid antibodies) or bruising within the last 12 months prior to consent.
14. Current or past cerebrovascular or cardiovascular disease or at risk of clotting disorders.
15. Impaired mobility (e.g., is wheelchair bound or bedridden) that, in the investigator's opinion, places the participant at increased risk of thrombosis.
16. Known or suspected carcinoma of the breast or suspected progestin-dependent neoplasia.
17. Known or suspected pelvic organ carcinoma.
18. Known Papanicolaou (Pap) or human papillomavirus (HPV) test abnormality that would require a repeat evaluation or treatment during study participation based on standard of care guidelines (American Society for Colposcopy and Cervical Pathology or American College of Obstetricians and Gynecologists).
19. Known benign or malignant liver tumors, renal disease, or active liver disease.
20. Invasive cancer (past history of any carcinoma or sarcoma, except non-melanoma skin cancer) unless in remission for >5 years.
21. Current or past medically diagnosed severe depression, which, in the investigator's opinion, could be exacerbated by use of a hormonal contraceptive, unless participant is on stable antidepressant medication.
22. Known or suspected current alcohol dependence syndrome or any recreational drug use that may affect metabolism of the IP or study compliance.
23. Abnormal screening laboratory values defined as:

    1. Fasting clinical chemistry values or CBC values designated clinically significant by the investigator.
    2. Liver function test results >twice the upper limit of normal.
24. Uncontrolled thyroid disorder.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 165 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the contraceptive efficacy of 2 LB SQ injections administered at a 4-month (approximately 17 weeks)interval over 8 cycles | 224 days
  As measured by The cumulative pregnancy percentage (calculated using Kaplan-Meier) through 8 cycles

SECONDARY OUTCOMES:
To assess the safety of 2 LB SQ injections | 240 days
  To assess the safety of 2 LB SQ injections as measured by:
  Number of participants with abnormal laboratory values and/or adverse events that are related to treatment
To further explore the contraceptive efficacy of 2 LB SQ injections | 224 days
  To further explore the contraceptive efficacy of 2 LB SQ injections as measured by the Pearl Index through 8 cycles
To explore bleeding patterns in participants receiving 2 LB SQ injections | 240 days
  To explore bleeding patterns in participants receiving 2 LB SQ injections as measured by Number of bleeding and spotting days per 30-, 90-, and 120-day intervals
To evaluate acceptability of 2 LB SQ injections | 240 days
  To evaluate acceptability of 2 LB SQ injections as measured by the number and percentage of subjects that provide each response to a given question related to acceptability on the CCN021b Acceptability and Satisfaction Questionnaire responses at 8 months.
  Questions range from 'Definitely No' to 'Definitely Yes'.
To evaluate satisfaction of 2 LB SQ injections | 240 days
  To evaluate satisfaction of 2 LB SQ injections as measured by the number and percentage of subjects that provide each response to a given question related to satisfaction on the CCN021b Acceptability and Satisfaction Questionnaire responses at 8 months.
  Questions range from 'Very Satisfied' to 'Very Unsatisfied' and 'Strongly Agree' to 'Strongly Disagree'.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, PhD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

IPD SHARING:
Plan to Share IPD: No